CLINICAL TRIAL: NCT06795334
Title: Long Term Impact of Induced Abortion: a Multicenter Prospective Cohort Study in China
Brief Title: Long Term Impact of Induced Abortion
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ChiCTR2400089586
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Non-medical Abortion Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Through prospective observation of the queue, the risks of mid to long term complications for Chinese women caused by surgical and medical abortion, as well as their potential impacts on women's fertility, pregnancy complications/comorbidities, and maternal and infant health, are identified. This provides scientific evidence for the assessment, protection, and preservation of fertility among Chinese women of childbearing age, and decision-making basis for the development and improvement of artificial abortion and fertility policies and guidelines for the country.

ELIGIBILITY:
Inclusion Criteria:

* Women who voluntarily request non-medical abortion surgery, early pregnancy (≤ 10 weeks of gestation); Age range: 20-40 years old (inclusive); Willingness to have another child; No long-term intention to go abroad during the research period; Willing to accept regular postoperative follow-up and voluntarily sign an informed consent form.

Exclusion Criteria:

* Pathological miscarriage such as spontaneous abortion and missed abortion; Difficulty in reading, writing, or understanding; Other situations deemed unsuitable for inclusion by doctors.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who voluntarily request non-medical abortion surgery, early pregnancy (≤ 10 weeks of gestation); Age range: 20-40 years old (inclusive); Willingness to have another child; No long-term intention to go abroad during the research period; Willing to accept regular postoperative follow-up and voluntarily sign an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
artificial abortion | 2 years

SECONDARY OUTCOMES:
medical abortion | 2 years

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR